CLINICAL TRIAL: NCT07168603
Title: A Phase I/II Clinical Trial to Evaluate Safety and Efficacy of Autologous Nucleus Pulposus Cells (aNPC) Transplantation in the Treatment of Degenerative Disc Disease
Brief Title: EvaluatIon of Autologous Nucleus Pulposus Cells (aNPC) in Degenerative Disc Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ASTEROGENE Biomedical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-001
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Intervertebral Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- aNPC will be injected into the degenerated disc to evaluate safety and efficacy (Experimental): Subjects will receive a single intradiscal injection of autologous nucleus pulposus cells (aNPC) into the degenerated central nucleus pulposus of the affected disc. The injection will be guided by C-arm X-ray to ensure accurate placement, and subjects will be followed for 12 months (52±2 weeks) for safety and efficacy assessments.
  Interventions: Drug: aNPC

INTERVENTIONS:
Drug: aNPC — Eligible subjects must be diagnosed with disc herniation and scheduled for discectomy, nucleus pulposus tissue will be collected for cell culture. Cultured cells will be then reintroduced into the degenerated disc via injection. Subjects will undergo multiple follow-up visits after surgery to evaluate safety and efficacy, supplemented with imaging studies to assess disc height, tissue regeneration, and water-retention capacity.
  Other Names: Autologous Nucleus Pulposus Cells

SUMMARY:
This is an open-label, single-center Phase I/II clinical trial investigating the safety and efficacy of autologous nucleus pulposus cells (aNPC) in patients with disc degeneration. Eligible participants are those assessed by the principal investigator to have disc herniation suitable for discectomy and confirmed disc degeneration. During the treatment period, participants will receive a single injection of autologous nucleus pulposus cells at a concentration of approximately 1×10⁶ viable cells/mL with a total volume not exceeding 3 mL. The injection will be guided by C-arm X-ray to ensure accurate placement into the degenerated central nucleus pulposus of the disc from which tissue was previously harvested. Participants will be followed for 12 months. Safety assessments will primarily include monitoring for inflammatory responses using ESR and CRP after cell injection, as well as recording any treatment-emergent adverse events (AEs). Efficacy will be evaluated using pain assessment and imaging outcomes, including lumbar X-ray and MRI reviewed independently by a radiologist. Additionally, patient-reported outcomes will assess quality of life improvements following treatment using the Visual Analogue Scale (VAS), Activities of Daily Living (ADLs), and the Oswestry Disability Index (ODI). Laboratory tests, including CBC/DC, BUN, creatinine, AST, and ALT, will also be conducted throughout the treatment and observation period to monitor participant safety.

DETAILED DESCRIPTION:
Degenerative disc disease (DDD) commonly occurs in adults and represents an irreversible aging process. It is also one of the primary causes of low-back pain (LBP). The nucleus pulposus possesses high water-retention capacity, allowing it to cushion the vertebrae and reduce friction during movement. However, with aging, the disc gradually loses its water absorption ability and becomes fibrotic, leading to structural degeneration. In addition, sports injuries or sudden mechanical stress may cause disc herniation, compressing spinal nerves and triggering both disc degeneration and back pain. The release of inflammatory mediators further induces severe pain. Once the nucleus pulposus herniates, the tissue continues to degenerate, placing greater stress on the surrounding annulus fibrosus. Over time, this accelerates the progression of DDD.

Regenerative medicine has recently emerged as a promising clinical treatment approach, aiming to restore or rebuild healthy tissue through biological means, with cell therapy being a key area of development. In our approach, autologous cells are harvested from patients' tissue, expanded and activated through ex vivo cell culture, and then reintroduced into the degenerated disc region under X-ray guidance. This autologous cell therapy avoids the risk of immune rejection or transplant-related complications. For patients undergoing treatment for disc herniation, discectomy not only relieves pain symptoms but also provides herniated disc tissue as an ideal source of autologous disc cells for further use in regenerative therapy. These cells can serve as a valuable implant material for disc repair.

The current clinical trial enrolls both male and female subjects aged ≥20 years who have not undergone prior disc surgery. Eligible patients must be diagnosed with disc herniation and scheduled for discectomy, during which nucleus pulposus tissue will be collected for cell culture. Following cell expansion, the cultured cells will be reintroduced into the degenerated disc region via injection. Subjects will undergo multiple follow-up visits within one year after surgery to evaluate safety and efficacy, supplemented with imaging studies to assess disc height, tissue regeneration, and water-retention capacity. Hence, the primary objective of this study is to evaluate the safety of aNPC during the treatment of disc degeneration. Secondary objectives include evaluating the effects of these cells on subjects' quality of life, as measured by Activities of Daily Living (ADLs) and the Oswestry Disability Index (ODI), on pain improvement assessed by the Visual Analogue Scale (VAS), and on imaging outcomes, including lumbar X-ray and MRI assessments, before and after treatment.

This clinical study will be conducted in accordance with the requirements of the Institutional Review Board (IRB) and will fully comply with Good Clinical Practice (GCP) standards and relevant regulations to minimize patient safety risks. In the future, this therapy has the potential to reduce the long-term reliance on pain medications, avoid associated side effects, slow disc degeneration, and alleviate pain and discomfort. Furthermore, it is expected to decrease the need for surgical interventions and provide a more effective and convenient therapeutic option for patients suffering from degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

* Main inclusion criteria:

  1. Age≧20 years old.
  2. Diagnosed with a disc herniation, can be having a discectomy.
  3. Having low back pain with affecting the lower limbs.
  4. Lower back pain should persist for more than six weeks and fail to improve with conservative treatments.
  5. VAS score ≥ 6.
  6. Single lumbar intervertebral disc degeneration or ruptured pinched nerve evaluated by Lumbar X-ray and MRI.
  7. Informed consent has been signed by subjects of his own accord.

Exclusion Criteria:

* 2. Main exclusion criteria:

  1. Levels of coagulation, liver, and kidney functions do not meet reference ranges. Following the reference range announced by the medical laboratory department at clinical trial institution, as shown below, PT/INR: 11-15 (sec)/ INR 0.78-1.12; BUN: 6.0-20.0 (mg/dL); Creatinine: (Female)0.5-0.9 (mg/dL)/ (Male)0.7-1.2 (mg/dL); AST (GOT): < 40 (U/L); ALT (GPT): < 41 (U/L)
  2. Bone marrow function did not meet specific criteria, including appropriate levels of white blood cells, platelets, and hemoglobin.

     Following the reference range announced by the medical laboratory department at clinical trial institution, as shown below, White blood cells: 4.00-11.00 (*103/μL); Platelets: 130-140 (*103/μL); Hemoglobin: Female: 12.0-16.0 (g/dL), Male: 13.0-17.0 (g/dL)
  3. Spinal inflammation, injury, or structural instability, including but not limited to the following：spondylodiscitis, spondylitis, spondylolisthesis, fracture, previous spinal trauma, severe spinal canal stenosis (hypertrophic fibrosis or ossification oof the ligamentum flavum), spinal tumor, metabolic bone disease.
  4. Local tissue infection or inflammation near the surgical site.
  5. Systemic infections require antibiotic treatment.
  6. Immunodeficiency disease or current use of immunosuppressive drugs.
  7. Tumor history.
  8. Severely degenerated or damaged annulus fibrosis, and the Pfirrman grade exceeds V.
  9. Hypersensitivity to penicillin, streptomycin, and amphotericin B or similar antibiotics.
  10. Cannot undergo discectomy.
  11. Autoimmune disease.
  12. Blood disease. (ex, anemia, blood coagulation dysfunction, leukemia, ITP, etc.)
  13. Spinal surgical treatment received.
  14. Drug allergy.
  15. Have been enrolled in other clinical trials in the past four weeks.
  16. Pregnancy and breastfeeding.
  17. Positive for HIV or VDRL in blood tests, as well as uncontrolled carriers of hepatitis B or C.
  18. Cannot take an MRI scan.
  19. Subjects who are not suitable for participating in this clinical trial diagnosed by PI.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
ESR: Erythrocyte Sedimentation Rate | From enrollment to the end of treatment at 52±2 weeks.
  A clinical test for detecting acute and chronic inflammation, representing non-specific tissue inflammation or damage. It will be measured to assess infectious inflammatory status, monitor disease progression, and evaluate treatment response.
  Unit of Measure: mm/hour
CRP: C-Reactive Protein | From enrollment to the end of treatment at 52±2 weeks.
  A specific protein which increases significantly during bacterial infections. It is a sensitive marker of inflammation and infection, responding more rapidly to changes in disease activity compared to ESR. CRP levels will be measured to assess inflammatory status and monitor therapeutic efficacy.
AE | From enrollment to the end of treatment at 52±2 weeks.
  Adverse events will be monitored and recorded for each participant from baseline through the treatment period. The relationship of each AE to the study treatment will be assessed. Severity and grading of AEs will follow the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0). Unit of Measure: Number and grade of AEs

SECONDARY OUTCOMES:
VAS: Visual Analogue Scale | From enrollment to the end of treatment at 52±2 weeks.
  VAS will be used to assessed pain intensity, which is a 10 cm line (0 to 10 cm) where 0 represents "no pain" and 10 represents "worst imaginable pain." Patients will mark their pain level on the scale, and the score will be recorded from.
  Unit of Measure: cm (0-10)
MRI | From enrollment to the end of treatment at 52±2 weeks.
  MRI will be used to evaluate tissue regeneration. Newly formed tissue appears as a deeper, more intense white signal on MRI images. Pre-treatment and post-treatment MRI images will be assessed by an independent radiology expert (not involved in the trial) to determine signal intensity, which will be used as a quantitative measure of tissue regeneration.
  Unit of Measure: Signal intensity
Lumbar X-ray | From enrollment to the end of treatment at 52±2 weeks.
  Lumbar X-rays will be used to assess disc degeneration. A decrease in disc height indicates degeneration. Disc height will be measured on pre-treatment and post-treatment X-ray images by independent evaluators, and the change will be used as a quantitative measure of treatment effect.
  Unit of Measure: mm
Quality of Life - Activities of Daily Living (ADLs) | From enrollment to the end of treatment at 52±2 weeks.
  ADLs will be assessed using a standardized questionnaire completed by each patient at each study visit. The scores from all items will be averaged to obtain a mean ADL score, which will serve as a reference for evaluating treatment effect on quality of life.
  Unit of Measure: Mean score (units on a scale)
Quality of Life - Oswestry Disability Index (ODI) | From enrollment to the end of treatment at 52±2 weeks.
  ODI：The ODI evaluates disability due to low back pain. It consists of 10 sections, each containing 6 statements scored from 0 to 5, with higher scores indicating greater disability. The total ODI score will be calculated pre-treatment and post-treatment to assess changes in patient disability.
  Unit of Measure: Total score (0-50)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) for this study. The primary reason is to protect participant privacy and confidentiality. In addition, institutional policy and applicable regulations do not permit release of raw participant-level data.